CLINICAL TRIAL: NCT05856383
Title: Efficacy and Safety of Inetetamab Combined With Pyrotinib and Vinorelbine in the Treatment of Advanced Breast Cancer
Brief Title: Efficacy and Safety of Inetetamab Combined With Pyrotinib and Vinorelbine in ABC
Acronym: HER2-VIP
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen Zhanhong, Clinical Professor, Zhejiang Cancer Hospital
Other Study IDs: ZCHBC024
Record Dates: First submitted 2023-04-02; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: HER2-positive Advanced Breast Cancer
Keywords: Advanced breast cancer，HER2-positive
MeSH Terms: interventions — pyrotinib; Vinorelbine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group of ues of inetetamab combined with pyrotinib and vinorelbine: Group of ues of inetetamab combined with pyrotinib and vinorelbine
  Interventions: Drug: Inetetamab Combined With Pyrotinib and Vinorelbine

INTERVENTIONS:
Drug: Inetetamab Combined With Pyrotinib and Vinorelbine — Inetetamab Combined With Pyrotinib and Vinorelbine

SUMMARY:
This is a prospective, no interventional, single arm cohort study, which aims to study the efficacy and safety of inetetamab combined with pyrotinib and vinorelbine in the Treatment of HER2 positive advanced breast cancer in the real world. The study will be conducted by signing an informed consent form for study enrollment, collecting patient case information, and conducting observation and follow-up.

DETAILED DESCRIPTION:
This is a prospective, no interventional, single arm cohort study, which aims to study the efficacy and safety of inetetamab combined with pyrotinib and vinorelbine in the Treatment of HER2 positive advanced breast cancer in the real world. The study will be conducted by signing an informed consent form for study enrollment, collecting patient case information, and conducting observation and follow-up.The research process is divided into screening period, treatment period, and survival and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. The HER2 positive advanced breast cancer confirmed by cytology or histology must meet the following conditions at the same time:

(1) HER2 positive is defined as>10% of immunoreactive cells with an immunohistochemical (IHC) score of 3 or an in situ hybridization (ISH) result of HER2 gene amplification (2) Advanced breast cancer is defined as locally advanced breast cancer or metastatic breast cancer that cannot be removed by radical surgery confirmed by researchers; 3. The functional level of the main organs has been evaluated by the researchers to withstand chemotherapy, anti HER2 monoclonal antibodies, and anti HER2 TKI drugs. The LVEF and QT intervals measured by echocardiography or MUGA are within a clinically acceptable safety range. If the survival benefits of the treatment value are assessed by the researcher to be greater than the risks faced, the admission conditions for the specific organ function level can be appropriately relaxed by the researcher, but the reasons need to be explained in the medical record; 4. ECOG score: 0-2 points; 5. Voluntarily sign the informed consent form for this study. 6. Contraception during the study period and within 6 months after treatment, non lactation.

Exclusion Criteria:

1. Pregnant or lactating women;
2. At the same time or in the past five years, patients with one or more malignant tumors with metastatic capacity or potential other than HER2 positive breast cancer, but not including cured cervical carcinoma in situ, thyroid cancer, skin basal cell carcinoma or squamous cell carcinoma. For other malignant tumors occurring within a period of more than 5 years from this treatment, if only cured by surgery, they are allowed to be included.
3. Persons with a known history of allergy to the drug components of this protocol;
4. Have a history of immunodeficiency, including HIV testing positive, or have other acquired or congenital immunodeficiency diseases;
5. The researcher believes that it is not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with HER2 positive dvanced breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progressive free survival(PFS) | From date of treatment of inetetamab combined with pyrotinib and vinorelbine until the date of the progression of the tumor or death from any cause, whichever came first, assessed up to about 48 months
  The time between the date of treatment of inetetamab combined with pyrotinib and vinorelbine and the progression of the tumor or death from any cause.
Adverse events | assessed up to 48 months
  The duration of adverse reaction data collection should be from the date the patient started medication to 30 days after the end of the last medication

SECONDARY OUTCOMES:
Overall Survival(OS) | From date of the patient starts treatment of inetetamab combined with pyrotinib and vinorelbine and vinorelbine and death from any cause，assessed up to about 48 months.
  Refers to the time between the date when the patient starts treatment of inetetamab combined with pyrotinib and vinorelbine and vinorelbine and death from any cause.
Objective response rate(ORR) | up to 48 months.
  Refers to the proportion of patients whose tumors have shrunk to a certain amount and remained for a certain period of time. The percentage of cases that include CR and PR in the number of evaluable cases.
Disease Control Rate (DCR) | up to 48 months.
  Refers to the percentage of confirmed cases of complete remission (CR), partial remission (PR), and disease stabilization (SD) (≥ 4 weeks) among patients with evaluable efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Chen zhanhong, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ma F, Ouyang Q, Li W, Jiang Z, Tong Z, Liu Y, Li H, Yu S, Feng J, Wang S, Hu X, Zou J, Zhu X, Xu B. Pyrotinib or Lapatinib Combined With Capecitabine in HER2-Positive Metastatic Breast Cancer With Prior Taxanes, Anthracyclines, and/or Trastuzumab: A Randomized, Phase II Study. J Clin Oncol. 2019 Oct 10;37(29):2610-2619. doi: 10.1200/JCO.19.00108. Epub 2019 Aug 20. PMID 31430226
- [Result] Xu B, Yan M, Ma F, Hu X, Feng J, Ouyang Q, Tong Z, Li H, Zhang Q, Sun T, Wang X, Yin Y, Cheng Y, Li W, Gu Y, Chen Q, Liu J, Cheng J, Geng C, Qin S, Wang S, Lu J, Shen K, Liu Q, Wang X, Wang H, Luo T, Yang J, Wu Y, Yu Z, Zhu X, Chen C, Zou J; PHOEBE Investigators. Pyrotinib plus capecitabine versus lapatinib plus capecitabine for the treatment of HER2-positive metastatic breast cancer (PHOEBE): a multicentre, open-label, randomised, controlled, phase 3 trial. Lancet Oncol. 2021 Mar;22(3):351-360. doi: 10.1016/S1470-2045(20)30702-6. Epub 2021 Feb 11. PMID 33581774